CLINICAL TRIAL: NCT02230020
Title: Efficacy of High Flow Therapy in COPD At Home
Acronym: EHFT
Status: Terminated | Type: Observational
Why Stopped: Sponsor funding
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: NA_00084508
Record Dates: First submitted 2014-08-29; First posted 2014-09-03 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — CRP Fibrinogen
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Nasal High Flow: All subjects are in this group
  Interventions: Device: Nasal High Flow

INTERVENTIONS:
Device: Nasal High Flow

SUMMARY:
Preliminary data show that in COPD patients, HFT substantially decreases ventilatory demand during sleep. The central hypothesis of this proposal is that lowering ventilatory demand using nasal high-flow therapy during sleep will elevate lung function, reduce dyspnea on exertion and improve quality of life. Thus, this proposal aims will determine the effects HFT over time on 1) lung function; 2) dyspnea on exertion; and 3) quality of life.

ELIGIBILITY:
Inclusion Criteria:

* 1. Consenting adults over the age of 18 with COPD

Exclusion Criteria:

* 1. Apnea Hypopnea Index>15 events/hr 2. Use of Non-invasive positive pressure ventilation (CPAP + Bilevel) 3. Severe bilateral nasal obstruction (apparent mouth breathing at rest) 4. Documented clinical cardiovascular disease, as defined below:

  1. myocardial infarction in past 3 months
  2. revascularization procedure in past 3 months
  3. implanted cardiac pacemaker or ICD
  4. unstable arrhythmias
  5. congestive heart failure with ejection fraction < 40%
  6. uncontrolled hypertension (BP > 190/110) 5. History of end stage renal disease (on dialysis) 6. History of end stage liver disease, such as:

  <!-- -->

  1. Jaundice
  2. ascites
  3. history of recurrent gastrointestinal bleeding
  4. transjugular intrahepatic portosystemic shunt (TIPS) ; 7. Transportation industry worker (commercial truck or bus drivers, airline pilots) 8. Known pregnancy (by self report) 9. Known coagulopathy or anticoagulant use (e.g. coumadin) other than aspirin. 10. Do you take medications for any of the following reasons:

  <!-- -->

  1. Pain control (besides NSAIDs)
  2. Sleep medication
  3. Benzodiazepines
  4. Methadone

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic Obstructive Pulmonary Disease
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2013-08-15 (Actual); Primary Completion 2015-12-13 (Actual); Study Completion 2015-12-13 (Actual)

PRIMARY OUTCOMES:
Lung Function | Baseline and 1 month
  Spirometry will be performed before and after each sleep study
Dyspnea score | Baseline and 1 month
  Borg scale score before and after each sleep study
Sleep quality | Baseline and 1 month
  Sleep architecture assessed from sleep studies
Quality of life | Baseline and 1 month
  St Georges Respiratory Questionnaire Hopkins Sleep Survey MRC Breathlessness Scale UCSD Shortness of Breath

CONTACTS AND LOCATIONS:
Overall Officials: Jason Kirkness, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States